CLINICAL TRIAL: NCT04785755
Title: Effects of Adding Hypertonic Saline Solutions and/or Etilefrine to Standard Diuretics Therapy in Egyptian Cirrhotic Patients With Ascites
Brief Title: Effects of Adding Hypertonic Saline Solutions and/or Etilefrine to Standard Diuretics Therapy in Hepatic Ascites
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hala Abd EL-Tawab Ibrahim Radwan (Other)
Responsible Party: Sponsor-Investigator, Hala Abd EL-Tawab Ibrahim Radwan, clinical pharmacy master degree, pharm D, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ascites of liver cirrhosis
Record Dates: First submitted 2021-02-26; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Hepatic Ascites
Keywords: Ascites, Hypertonic saline, Etilefrine, Aldosterone, Leptin.
MeSH Terms: conditions — Ascites | interventions — Furosemide; Spironolactone; Saline Solution, Hypertonic; Sodium Chloride; Etilefrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Active Comparator): The control group (n=15) received oral standard diuretic therapy (furosemide 40 mg tablet plus spironolactone 100 mg tablet with a dose increase in 40 mg:100 mg ratio) given once daily in the morning for 38 days (from the first day of the study to the end of the study).
  Interventions: Drug: Oral standard diuretics therapy
- Group II (Experimental): The hypertonic saline solution (HSS) group (n=25) received oral standard diuretic therapy (furosemide 40 mg tablet plus spironolactone 100 mg tablet with a dose increase in 40 mg:100 mg ratio) given once daily in the morning for 38 days (from the start of the study to the end of the study) with hypertonic saline solution (150ml, 1.4% - 4.6%) infused slowly over one hour peripherally once daily from the first day of the study for eight days.
  Interventions: Drug: Oral standard diuretics therapy; Drug: Hypertonic saline solution
- Group III (Experimental): The etilefrine group (n=25) received oral standard diuretic therapy (furosemide 40 mg tablet plus spironolactone 100 mg tablet with a dose increase in 40 mg:100 mg ratio) given once daily in the morning for 38 days (from the first day of the study to the end of the study), and etilefrine 5 mg tablet given by mouth three times daily for 38 days (from the first day of the study to the end of the study).
  Interventions: Drug: Oral standard diuretics therapy; Drug: Etilefrine
- Group IV (Experimental): The hypertonic saline solution (HSS) + Etilefrine group (n=25) received oral standard diuretic therapy (furosemide 40 mg tablet plus spironolactone 100 mg tablet with a dose increase in 40 mg100mg ratio) given once daily in the morning for 38 days (from the first day of the study to the end of the study), with hypertonic saline solution (150ml, 1.4% - 4.6%) infused slowly over one hour peripherally once daily from the first day of the study for eight days, and etilefrine 5 mg tablet given by mouth three times daily for 38 days (from the first day of the study to the end of the study).
  Interventions: Drug: Oral standard diuretics therapy; Drug: Hypertonic saline solution; Drug: Etilefrine

INTERVENTIONS:
Drug: Oral standard diuretics therapy — Oral standard diuretics therapy (furosemide 40 mg tablet plus spironolactone 100 mg tablet with a dose increase in 40 mg:100 mg ratio) given once daily in the morning for 38 days (from the first day of the study to the end of the study).
  Other Names: Furosemide (lasix®), Spironolactone (Aldactone®)
Drug: Hypertonic saline solution — Hypertonic saline solution (150ml, 1.4% - 4.6%) infused slowly over one hour peripherally once daily from the first day of the study for eight days.
  Other Names: prepared from sodium chloride 0.9% intravenous solution and sodium chloride 3% intravenous solution (, Egypt Otsuka Pharmaceutical Co.).
  Arms: Group II; Group IV
Drug: Etilefrine — Etilefrine 5 mg tablet given by mouth three times daily for 38 days (from the first day of the study to the end of the study).
  Other Names: (Vascon®)
  Arms: Group III; Group IV

SUMMARY:
This work aimed to evaluate and compare the impact of adding hypertonic saline solution (HSS) infusion and/or etilefrine to oral diuretics therapy on clinical outcomes, renal and systemic hemodynamics, metabolic and inflammatory pathways by estimating the changes in selected biological markers in cirrhotic patients with ascites. Also, the trial aims to assess the safety and tolerability of such treatment regimens.

DETAILED DESCRIPTION:
This comparative, randomized, prospective controlled clinical trial was conducted on 90 cirrhotic patients with ascites who were admitted to the Hepatology Department of National Liver Institute, Menoufiya University. The study was approved by the Institution Review Board (IRB) of the National Liver Institute (NLI), Menoufiya University, Egypt with NLI/IRB protocol number: 00131/2017. Informed consent was obtained from all patients who participated in the study.

Patients were randomized into four groups:

Group I: (n=15) received oral standard diuretic therapy (furosemide 40 mg plus spironolactone 100 mg with dose increase in 40 mg :100 mg ratio).

Group II: (n=25) received (150 ml,1.4% - 4.6%) of hypertonic saline solution (HSS) plus standard diuretics therapy.

Group III: (n=25) received etilefrine 5 mg tablets 3 times daily plus standard diuretics therapy.

Group IV: (n=25) received (150 ml, 1.4% - 4.6%) of HSS and etilefrine 5 mg tablets 3 times daily plus standard diuretics therapy.

Time frame:

Oral standard diuretics therapy administered for 38 days. Etilefrine tablets administered for 38 days. Infusion of HSS administered for eight days. Diuretics dosage reassessed according to blood pressure, diuresis, serum sodium, and serum potassium levels.

All blood and urine samples were collected and measured as follows:

1. At baseline before initiation of any treatment (first measurement)
2. Eight days after treatment with studied medications (second measurement).
3. One month after the second measurement (third measurement).

Samples collection:

Venous blood samples were drawn from enrolled patients in the morning before treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement). Blood samples were centrifuged and the resulting supernatant was frozen at -80 C until all samples were collected. 24-hr urine was collected in the morning from 7 am to 7 am of the next day before initiation of treatment, after eight days of treatment, and after a month from the second measurement to assess diuresis and urinary creatinine, urinary Na, and urinary K, also hepatic and renal functions, complete blood count, serum levels of c-reactive protein, interleukin-6, aldosterone, and leptin were measured at baseline, after eight days and, after a month from the second measurement.

ELIGIBILITY:
Inclusion Criteria:

* All cirrhotic patients with ascites grade I- III.
* Patients ages from 25 -65 years.

Exclusion Criteria:

* Non-cirrhotic ascites.
* Congestive heart failure.
* Acute renal failure.
* Hepatocellular carcinoma.
* All Cancer types.
* Arterial hypertension.
* Acute infection.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluate and compare the impact of adding hypertonic saline solution (HSS) infusion and/or etilefrine to oral standard diuretics therapy on the inflammatory pathway in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in serum interleukin-6 (pg/ml) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected for measuring from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the impact of adding HSS infusion and/or etilefrine to oral standard diuretics therapy on the serum C-reactive protein in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in serum C-reactive protein (mg/L) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected for measuring from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to the standard oral standard diuretics therapy on the metabolic pathway in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in serum leptin (pg/ml) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected for measuring from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the impact of adding HSS solution infusion and/or etilefrine to oral standard diuretics therapy on the renal hemodynamics in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in plasma aldosterone (pg/ml) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected for measuring from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the impact of adding HSS infusion and/or etilefrine to oral diuretics therapy on the diuresis of cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in 24-hour urine output (ml/24 hr) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). 24-hr urine was collected in the morning from 7 am to 7 am of the next day before treatment (first collection), after eight days of treatment (second collection), and after a month from the second collection for assessing diuresis.
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to oral diuretics therapy on the systemic hemodynamic of cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the effects of the treatments on mean arterial pressure (MAP) in patients with ascites. Systolic blood pressure (mmHg) and diastolic blood pressure (mmHg) were measured using a sphygmomanometer to calculate MAP first on day one of the treatments (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement). Final changes in MAP (mmHg) were calculated from the first day of the study to the end of the study (study duration 38 days)
Evaluate the effect of adding HSS infusion and/or etilefrine to oral diuretics therapy on serum sodium (Na) concentration in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in serum Na concentration (mEq/L) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate the effect of adding HSS infusion and/or etilefrine to oral diuretics therapy on serum creatinine concentration in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in serum creatinine concentration (mg/dl) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected for measuring from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).

SECONDARY OUTCOMES:
Evaluate the effect of adding HSS infusion and/or etilefrine to oral diuretics therapy on prothrombin concentration in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in prothrombin concentration (%) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to oral diuretics therapy on the model of end-stage liver disease (MELD score)in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By calculating the final change in MELD score in patients with ascites to assess the severity of liver disease for transplant planning, from the first day of the study to the end of the study (study duration 38 days). MELD score calculation depends on serum creatinine, serum bilirubin, prothrombin time, and the score calculated by a suitable online medical calculator. All blood samples were collected for measuring from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to the standard oral diuretics therapy on the model of end-stage liver disease depending on sodium (MELD score-Na)in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By calculating the final change in MELD-Na score in patients with ascites from the first day of the study to the end of the study (study duration 38 days). MELD-Na score calculation depends on serum creatinine, serum bilirubin, serum Na, prothrombin time, and the score calculated by a suitable online medical calculator. All blood samples were collected for measuring from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to oral diuretics therapy on Child-Pugh score in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By calculating the final change in Child-Pugh score in patients with ascites to assess the prognosis in liver cirrhosis from the first day of the study to the end of the study (study duration 38 days). Child-Pugh score calculation depends on serum albumin, serum bilirubin, prothrombin time, ascites, and encephalopathy grades. The score was calculated by a suitable online medical calculator. All blood samples were collected for measuring from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to the standard oral diuretics therapy on the bodyweight in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By calculating the final change in the patients' weight (kg) from the first day of the study to the end of the study (study duration 38 days). All enrolled patients were weighed by suitable weight scale on the morning of the first day of the study (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to the standard oral diuretics therapy on urinary sodium excretion in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in urinary Na concentration (mEq/24 hr) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). Urinary Na concentration was measured from a 24-hr urine collection sample. 24-hr urine was collected in the morning from 7 am to 7 am of the next day before initiation of the treatment (first measurement), after eight days of the treatment (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to the standard oral diuretics therapy on urinary creatinine excretion in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in urinary creatinine concentration (mg/dl) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). 24-hr urine collected in the morning from 7 AM to 7 AM of the next day before initiation of the study to measure urinary creatinine concentration (first measurement), after eight days of treatment (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to the standard oral diuretics therapy on serum alanine aminotransferase enzyme (ALT) in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in serum ALT (U/L) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to the standard oral diuretics therapy on serum albumin in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in serum albumin (mg/dl) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to the standard oral diuretics therapy on serum total bilirubin in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in serum total bilirubin (mg/dl) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to the standard oral diuretics therapy on serum blood urea nitrogen (BUN) in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in serum BUN (mg/dl) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).
Evaluate and compare the effect of adding HSS infusion and/or etilefrine to the standard oral diuretics therapy on hemoglobin concentration in cirrhotic patients with ascites. | 38 days (from the first day of the study to the end of the study)
  By measuring the final change in hemoglobin concentration (gm/dl) in patients with ascites from the first day of the study to the end of the study (study duration 38 days). All blood samples were collected from enrolled patients in the morning on the first day of treatment (first measurement), after eight days (second measurement), and after a month from the second measurement (third measurement).

OTHER OUTCOMES:
Safety of adding HSS infusion and/or etilefrine to the standard oral diuretics therapy in cirrhotic patients with ascites. | 38 days (from the start of the study to the end of the study).
  Assessed by the number of patients who developed any new episodes of spontaneous bacterial peritonitis (SBP), new onset of hepatic encephalopathy (HE), the incidence of gastrointestinal bleeding, the incidence of hepatorenal syndrome (HRS), or renal impairment (increase in serum creatinine > 50% above the baseline. All assessments of enrolled patients were reported in the safety sheets.
Tolerability of adding HSS infusion and/or etilefrine to the standard oral diuretics therapy in cirrhotic patients with ascites. | 38 days (from the start of the study to the end of the study).
  Assessed by the number of patients who developed any unwanted side effects were reported from the treatment regimen as osmotic demyelination syndrome (ODS), vein extravasation, hypokalemia, acute hypotension, and laboratory abnormalities. All assessments of enrolled patients were reported in tolerability sheets.

CONTACTS AND LOCATIONS:
Overall Officials: Gamal A Badra, professor, Study Director — national liver institute / menoufiya university; Sahar El-Haggar, professor, Study Director — Tanta University; hala El said, professor, Study Director — national liver institute / menoufiya university
Locations (1):
- National liver institute- menoufiya university, Shibīn al Kawm, Monufia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reynolds TB. Ascites. Clin Liver Dis. 2000 Feb;4(1):151-68, vii. doi: 10.1016/s1089-3261(05)70101-x. PMID 11232182
- [Result] Gu XB, Yang XJ, Zhu HY, Xu BY. Effect of a diet with unrestricted sodium on ascites in patients with hepatic cirrhosis. Gut Liver. 2012 Jul;6(3):355-61. doi: 10.5009/gnl.2012.6.3.355. Epub 2012 Jul 12. PMID 22844565
- [Result] Morando F, Rosi S, Gola E, Nardi M, Piano S, Fasolato S, Stanco M, Cavallin M, Romano A, Sticca A, Caregaro L, Gatta A, Angeli P. Adherence to a moderate sodium restriction diet in outpatients with cirrhosis and ascites: a real-life cross-sectional study. Liver Int. 2015 May;35(5):1508-15. doi: 10.1111/liv.12583. Epub 2014 May 21. PMID 24811138
- [Result] Sam J, Nguyen GC. Protein-calorie malnutrition as a prognostic indicator of mortality among patients hospitalized with cirrhosis and portal hypertension. Liver Int. 2009 Oct;29(9):1396-402. doi: 10.1111/j.1478-3231.2009.02077.x. Epub 2009 Jul 7. PMID 19602136
- [Result] Eghtesad S, Poustchi H, Malekzadeh R. Malnutrition in liver cirrhosis:the influence of protein and sodium. Middle East J Dig Dis. 2013 Apr;5(2):65-75. PMID 24829672
- [Result] Arroyo V, Fernandez J. Relationship between systemic hemodynamics, renal dysfunction, and fluid retention in cirrhosis. Clin Liver Dis (Hoboken). 2013 Jun 21;2(3):120-122. doi: 10.1002/cld.185. eCollection 2013 Jun. No abstract available. PMID 30992841
- [Result] Guo TT, Yang Y, Song Y, Ren Y, Liu ZX, Cheng G. Effects of midodrine in patients with ascites due to cirrhosis: Systematic review and meta-analysis. J Dig Dis. 2016 Jan;17(1):11-9. doi: 10.1111/1751-2980.12304. PMID 26630543
- [Result] Singh V, Dhungana SP, Singh B, Vijayverghia R, Nain CK, Sharma N, Bhalla A, Gupta PK. Midodrine in patients with cirrhosis and refractory or recurrent ascites: a randomized pilot study. J Hepatol. 2012 Feb;56(2):348-54. doi: 10.1016/j.jhep.2011.04.027. Epub 2011 Jul 13. PMID 21749847
- [Result] Hatanaka E, Shimomi FM, Curi R, Campa A. Sodium chloride inhibits cytokine production by lipopolysaccharide-stimulated human neutrophils and mononuclear cells. Shock. 2007 Jan;27(1):32-5. doi: 10.1097/01.shk.0000238061.69579.a5. PMID 17172977
- [Result] Kolsen-Petersen JA. Immune effect of hypertonic saline: fact or fiction? Acta Anaesthesiol Scand. 2004 Jul;48(6):667-78. doi: 10.1111/j.1399-6576.2004.00396.x. PMID 15196097
- [Result] Perez-Perez A, Vilarino-Garcia T, Fernandez-Riejos P, Martin-Gonzalez J, Segura-Egea JJ, Sanchez-Margalet V. Role of leptin as a link between metabolism and the immune system. Cytokine Growth Factor Rev. 2017 Jun;35:71-84. doi: 10.1016/j.cytogfr.2017.03.001. Epub 2017 Mar 4. PMID 28285098
- [Result] Buechler C, Haberl EM, Rein-Fischboeck L, Aslanidis C. Adipokines in Liver Cirrhosis. Int J Mol Sci. 2017 Jun 29;18(7):1392. doi: 10.3390/ijms18071392. PMID 28661458
- [Result] Reynolds TB, Lieberman FL, Goodman AR. Advantages of treatment of ascites without sodium restriction and without complete removal of excess fluid. Gut. 1978 Jun;19(6):549-53. doi: 10.1136/gut.19.6.549. PMID 680588
- [Result] Lafreniere G, Beliveau P, Begin JY, Simonyan D, Cote S, Gaudreault V, Israeli Z, Lavi S, Bagur R. Effects of hypertonic saline solution on body weight and serum creatinine in patients with acute decompensated heart failure. World J Cardiol. 2017 Aug 26;9(8):685-692. doi: 10.4330/wjc.v9.i8.685. PMID 28932357
- [Result] Henriksen JH, Fuglsang S, Bendtsen F, Moller S. Arterial hypertension in cirrhosis: arterial compliance, volume distribution, and central haemodynamics. Gut. 2006 Mar;55(3):380-7. doi: 10.1136/gut.2005.064329. PMID 16474108
- [Result] Li H, Guo Z, Yang X, Sun D. Mean arterial pressure drop is an independent risk factor of death in patients with HBV-related cirrhosis ascites. Turk J Gastroenterol. 2017 Jan;28(1):26-30. doi: 10.5152/tjg.2016.0412. Epub 2016 Dec 19. PMID 27991854
- [Result] Drazner MH, Palmer BF. Hypertonic saline: a novel therapy for advanced heart failure? Am Heart J. 2003 Mar;145(3):377-9. doi: 10.1067/mhj.2003.165. No abstract available. PMID 12660656
- [Result] Tuttolomondo A, Di Raimondo D, Bellia C, Clemente G, Pecoraro R, Maida C, Simonetta I, Vassallo V, Di Bona D, Gulotta E, Ciaccio M, Pinto A. Immune-Inflammatory and Metabolic Effects of High Dose Furosemide plus Hypertonic Saline Solution (HSS) Treatment in Cirrhotic Subjects with Refractory Ascites. PLoS One. 2016 Dec 12;11(12):e0165443. doi: 10.1371/journal.pone.0165443. eCollection 2016. PMID 27941973
- [Result] Okuhara Y, Hirotani S, Naito Y, Nakabo A, Iwasaku T, Eguchi A, Morisawa D, Ando T, Sawada H, Manabe E, Masuyama T. Intravenous salt supplementation with low-dose furosemide for treatment of acute decompensated heart failure. J Card Fail. 2014 May;20(5):295-301. doi: 10.1016/j.cardfail.2014.01.012. Epub 2014 Jan 22. PMID 24462960
- [Result] Haberl J, Zollner G, Fickert P, Stadlbauer V. To salt or not to salt?-That is the question in cirrhosis. Liver Int. 2018 Jul;38(7):1148-1159. doi: 10.1111/liv.13750. Epub 2018 May 16. PMID 29608812
- [Result] Tuttolomondo A, Pinto A, Di Raimondo D, Corrao S, Di Sciacca R, Scaglione R, Caruso C, Licata G. Changes in natriuretic peptide and cytokine plasma levels in patients with heart failure, after treatment with high dose of furosemide plus hypertonic saline solution (HSS) and after a saline loading. Nutr Metab Cardiovasc Dis. 2011 May;21(5):372-9. doi: 10.1016/j.numecd.2009.10.014. Epub 2010 Mar 25. PMID 20346637
- [Result] Gauthier A, Levy VG, Quinton A, Michel H, Rueff B, Descos L, Durbec JP, Fermanian J, Lancrenon S. Salt or no salt in the treatment of cirrhotic ascites: a randomised study. Gut. 1986 Jun;27(6):705-9. doi: 10.1136/gut.27.6.705. PMID 3522371